CLINICAL TRIAL: NCT00129623
Title: Double-blind, Placebo-controlled, Randomized, Multicenter Study to Assess the Efficacy and Safety of Oral Ibandronate Once Monthly in Postmenopausal Women With Osteopenia
Brief Title: A Study of Bonviva (Ibandronate) Once Monthly in Post-Menopausal Women With Osteopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BA18492
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Post-Menopausal Osteopenia
MeSH Terms: interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po monthly for 1 year
  Arms: 2
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 1 year
  Arms: 1

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of oral Bonviva 150mg once monthly compared with placebo in post-menopausal women with osteopenia. Patients will be randomized to receive either Bonviva 150mg po monthly, or placebo monthly. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* women 45-60 years of age;
* post-menopausal;
* ambulatory.

Exclusion Criteria:

* vertebral fracture (except traumatic fracture such as in a motor vehicle accident);
* low-trauma osteoporotic fracture in any other bone;
* breast cancer diagnosed within last 20 years;
* other malignancy diagnosed within last 10 years, except successfully resected basal cell cancer;
* treatment with any bisphosphonate within last 2 years;
* treatment with other drugs affecting bone metabolism within last 6 months.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (12):
  - Lakewood, Colorado
  - Stuart, Florida
  - Bethesda, Maryland
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Cincinnati, Ohio
  - Portland, Oregon
  - Amarillo, Texas
  - Norfolk, Virginia
  - Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in the United States.
Pre-assignment Details: Of the 451 participants who were screened, 160 participants were randomly assigned to the two treatment arms (Placebo and Ibandronate). The major reason for screening failure was participants did not meet the Bone Mineral Density (BMD) entry criteria.
Groups:
- Placebo: Participants with postmenopausal osteopenia were administered matching placebo tablet orally once monthly. All participants received OSCAL tablet (containing 500 mg calcium and 400 international units [IU] vitamin D) once a day as dietary supplements for the duration of the study. Participants received a total of 12 months of treatment and were followed for an additional period of 15 days.
- Ibandronate (IBN) 150 mg Monthly: Participants with postmenopausal osteopenia were administered 150 mg Ibandronate (IBN) tablet orally once monthly. All participants received OSCAL tablet (containing 500 mg/d calcium and 400 international units [IU]/d vitamin D) once a day as dietary supplements, for the duration of the study. Participants received a total of 12 months of treatment and were followed for an additional period of 15 days.
Period: Overall Study
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Started | 83 | 77
Intent-to-treat (ITT)/ Safety Population | 83 | 77
Completed | 73 | 65
Not Completed | 10 | 12
Not completed — Adverse Event | 3 | 7
Not completed — Refused Treatment | 5 | 3
Not completed — Failure to Return | 1 | 1
Not completed — Relocated job out of state | 1 | 0
Not completed — Uncertainty to return | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the safety population which included participants who had at least one dose of the trial medication documented in the case report form (CRF) whether withdrawn prematurely or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly | Total
Number analyzed (Participants) | 83 | 77 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (3.83) | 53.7 (3.64) | 53.5 (3.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 77 | 160
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Mean Bone Mineral Density (BMD) of the Lumbar Spine (L2 to L4) at Month 12
Description: BMD was measured by a single dual-energy x-ray absorptiometry (DEXA) scan of the lumbar spine at the time of screening and at Month 12. A BMD measurement was considered unsuitable in case of detection of a fracture, an osteoarthritic process, or a scanning artifact that could not be removed to such a degree that accurate measurement of BMD would be considered jeopardized by the central reading center. The change in BMD was defined as the relative difference between the last individual measurement available at 12 months and Baseline, using the following formula: Relative change = 100 x (BMD at 1 year - BMD at baseline) / (BMD at baseline)
Time Frame: Baseline and Month 12
Population: The ITT population included participants who were randomized, received at least one dose of the trial medication and had baseline and at least one follow-up evaluation data point.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 70 | 68
Percentage | -0.3941 (0.4148) | 3.7285 (0.4229)
Statistical Analysis 1: Comparison: Placebo vs Ibandronate (IBN) 150 mg Monthly; H0 (null hypothesis): There was no statistically significant difference between monthly treatment with 150 mg oral IBN and monthly treatment with placebo in relative change from baseline of mean lumbar spine (L2-L4 BMD). H1 (alternative hypothesis): There was a statistically significant difference between monthly treatment with 150 mg oral IBN and monthly treatment with placebo in relative change from baseline of mean lumbar spine (L2-L4 BMD); Test type: Superiority or Other; p < 0.0001, ANOVA — The primary analysis was an ANOVA (two way classification), including treatment group and time since menopause (as a binary variable; 0.5-3 years, >3 years) as independent factors; Mean Difference (Net) = 4.1226, 95% CI 2-sided [2.9613 to 5.2838]

2. Secondary Outcome: Absolute Change From Baseline in Mean Lumbar Spine BMD at Month 12
Description: BMD was measured by a single dual-energy x-ray absorptiometry (DEXA) scan of the lumbar spine at the time of screening and at Month 12. A BMD measurement was considered unsuitable in case of detection of a fracture, an osteoarthritic process, or a scanning artifact that could not be removed to such a degree that accurate measurement of BMD would be considered jeopardized by the central reading center. The absolute change from Baseline in mean BMD of the lumbar spine (L2-L4) was measured as g/cm^2 and summarized using descriptive statistics.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 70 | 68
g/cm^2 | -0.0039 (0.0319) | 0.0322 (0.0315)

3. Secondary Outcome: Relative Change From Baseline in Mean Proximal Femur BMD at Month 12
Description: BMD was measured by a single DEXA scan of the proximal femur at the time of screening and at Month 12. The relative (%) change from Baseline in BMD of the proximal femur (total hip, trochanter, femoral neck) at Month 12 was summarized using descriptive statistics. BMD of fractured bones that could impact the scan area were not taken into account.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 71 | 68
Percentage
  Total hip | -0.9265 (1.8790) | 1.4855 (2.1862)
  Trochanter | -0.9120 (3.0025) | 2.8688 (3.0906)
  Femoral Neck | -0.7537 (3.7743) | 1.0930 (2.6466)

4. Secondary Outcome: Absolute Change From Baseline in BMD of the Proximal Femur at Month 12
Description: BMD was measured by a single DEXA scan of the proximal femur at the time of screening and at Month 12. The absolute change from baseline in BMD of the proximal femur (total hip, trochanter, femoral neck) at Month 12 was summarized using descriptive statistics. BMD of fractured bones that could impact the scan area were not taken into account.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 71 | 68
g/cm^2
  Total hip | -0.0083 (0.0163) | 0.0133 (0.0194)
  Trochanter | -0.0061 (0.0185) | 0.0182 (0.0199)
  Femoral neck | -0.0061 (0.0284) | 0.0078 (0.0202)

5. Secondary Outcome: Relative Change From Baseline in Serum C-telopeptide Crosslinks of Type 1 Collagen (CTX)
Description: Fasting blood samples were collected from participants for analysis of serum CTX (sCTX), which is a biochemical marker of bone resorption. Relative change from baseline of sCTX after 3, 6, and 12 months of treatment was summarized using descriptive statistics.
Time Frame: Baseline and 3, 6 and 12 months
Population: The ITT population included participants who were randomized, received at least one dose of the trial medication and had baseline and at least one follow-up evaluation data point. n = the number of participants analyzed at a given time point.
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 83 | 77
Percentage
  Month 3, n = 81, 72 | -4.2230 [-11.4068 to 2.2989] | -55.7688 [-61.9565 to -46.7669]
  Month 6, n = 77, 72 | -6.5934 [-14.3590 to 0.6658] | -61.6459 [-64.5652 to -52.3364]
  Month 12, n = 75, 68 | -6.7416 [-14.6388 to 5.9238] | -56.5432 [-61.8357 to -46.7836]

6. Secondary Outcome: Absolute Change From Baseline in sCTX
Description: Fasting blood samples were collected from participants for analysis of sCTX, which is a biochemical marker of bone resorption. Absolute change from baseline of sCTX after 3, 6, and 12 months of treatment was summarized using descriptive statistics.
Time Frame: Baseline and 3, 6, 12 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: ng/ml
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 83 | 77
ng/ml
  Month 3, n = 81, 72 | -0.0350 [-0.0620 to 0.0130] | -0.2570 [-0.2930 to -0.2060]
  Month 6, n = 77, 72 | -0.0350 [-0.0670 to 0.0050] | -0.2675 [-0.3090 to -0.2300]
  Month 12, n = 75, 68 | -0.0320 [-0.0890 to 0.0250] | -0.2560 [-0.3030 to -0.1850]

7. Secondary Outcome: Percentage of Responders
Description: Percent responders were defined as follows: Participants with a) lumbar spine (LS) BMD, equal to or above Baseline at Month 12 b) proximal femur BMD, equal to or above Baseline at Month 12 c) Both lumbar spine and proximal femur BMD, equal or above Baseline at Month 12. BMD of the lumbar spine was defined as the BMD of at least two vertebrae (L2-L4) that were not fractured and not affected by an osteoarthritic process, or a scanning artifact that could not be removed to such a degree that accurate measurement of BMD would be considered jeopardized by the central reading center. Proximal femur included total hip, trochanter and femoral neck sites.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage
Groups:
- Placebo: Participants with postmenopausal osteopenia who were administered matching placebo tablet PO once monthly. All participants received 500 mg/d calcium and 400 international units [IU]/d vitamin D as dietary supplements consisting of one tablet a day of OSCAL for the duration of the study. Participants received 12 months of treatment and were followed for an additional period of 15 days.
- Ibandronate (IBN) 150 mg Monthly: Participants with postmenopausal osteopenia who were administered 150 mg IBN tablet orally (PO) once monthly. All participants received 500 mg/d calcium and 400 international units [IU]/d vitamin D as dietary supplements consisting of one tablet a day of OSCAL for the duration of the study. Participants received 12 months of treatment and were followed for an additional period of 15 days.
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 83 | 77
Percentage
  Lumbar spine equal to or above baseline | 38.6 | 88.2
  Proximal femur equal to or above baseline | 15.5 | 60.3
  LS and proximal femur equal to or above baseline | 8.5 | 54.4
Statistical Analysis 1: Comparison: Placebo vs Ibandronate (IBN) 150 mg Monthly; Lumbar BMD: Adjusted treatment effect - The treatment effect and 95% C.I. were represented by presenting OR. These were estimated by fitting a logistic regression model, with responder outcome (responder/non-responder) as the dependent variable and the treatment group (oral IBN 150 mg/Placebo) and time since menopause as the independent variables. An OR of >1 indicated participants treated with IBN were more likely to have BMD above or equal to baseline relative to those treated with placebo; Test type: Superiority or Other; Odds Ratio (OR) = 12.51, 95% CI 2-sided [5.12 to 30.56]
Statistical Analysis 2: Comparison: Placebo vs Ibandronate (IBN) 150 mg Monthly; Proximal femur BMD: The adjusted treatment effect and 95% C.I. were represented by presenting OR. These were estimated by fitting a logistic regression model, with responder outcome (responder/non-responder) as the dependent variable and the treatment group (oral IBN 150 mg once monthly/Placebo) and time since menopause as the independent variables. An OR of >1 indicated participants treated with IBN were more likely to have BMD above or equal to baseline relative to those treated with placebo; Test type: Superiority or Other; Odds Ratio (OR) = 8.59, 95% CI 2-sided [3.80 to 19.42]
Statistical Analysis 3: Comparison: Placebo vs Ibandronate (IBN) 150 mg Monthly; Lumbar Spine and Proximal Femur BMD: The adjusted treatment effect and 95% C.I. were represented by presenting OR. These were estimated by fitting a logistic regression model, with responder outcome (responder/non-responder) as the dependent variable, and treatment group (oral IBN150 mg/Placebo) and time since menopause as the independent variables. An OR of >1 indicated participants treated with IBN were more likely to have BMD above or equal to baseline relative to those treated with placebo; Test type: Superiority or Other; Odds Ratio (OR) = 13.80, 95% CI 2-sided [5.17 to 36.79]

8. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to 15 days after end of study treatment (Approximately 2 years)
Population: The safety population included participants who had at least one dose of the trial medication documented in the CRF whether withdrawn prematurely or not.
Measure: Number; unit: participants
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 83 | 77
participants
  Any AE | 64 | 60
  SAE | 1 | 3

9. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Blood for laboratory tests was taken at screening and immediately before participants received their monthly study medication at months 3, 6, and 12. The laboratory tests included: Hematology [white blood cells (WBCs), platelets, hematocrit, and hemoglobin] and Chemistry [albumin, creatinine, blood urea nitrogen (BUN), alanine aminotransferase (ALT), total calcium, 25-hydroxy vitamin D, phosphate, magnesium, sodium, potassium, and chloride].
Time Frame: Screening up to 12 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Number analyzed (Participants) | 83 | 77
participants
  WBC, low | 1 | 0
  ALT, high | 2 | 0
  Phosphate, high | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 days after end of study treatment (Approximately 2 years)
Description: SAEs and non-serious AEs were reported for members of the safety population, comprised of participants who had at least one dose of the trial medication documented in the CRF whether withdrawn prematurely or not.
Arm/Group | Placebo | Ibandronate (IBN) 150 mg Monthly
Serious Adverse Events (participants affected / at risk) | 1/83 | 3/77
Other Adverse Events (participants affected / at risk) | 41/82 | 40/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Ibandronate (IBN) 150 mg Monthly (N=77)
Cellulitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Chest pain (General disorders) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Ibandronate (IBN) 150 mg Monthly (N=76)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 12 | 6
Nasopharyngitis (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 5
Dental caries (Gastrointestinal disorders) | 3 | 4
Depression (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 4
Headache (Nervous system disorders) | 4 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4
Influenza like illness (General disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.